CLINICAL TRIAL: NCT05821361
Title: Hepatic Arterial Infusion of Oxaliplatin Plus Fluorouracil/Leucovorin Combined With Cadonilimab and Bevacizumab as First-line Therapy in Unresectable Hepatocellular Carcinoma: a Single Center, Open Label, Single Arm,, Phase II Trial
Brief Title: HAIC Combined With Cadonilimab and Bevacizumab as First-line Therapy in Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, HuiKai Li, Professor and Chief Surgeon, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N-0052
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Unrescetable Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+cadonilimab+bev (Experimental)
  Interventions: Drug: HAIC+Cadonilimab+Bevacizumab

INTERVENTIONS:
Drug: HAIC+Cadonilimab+Bevacizumab — Cadonilimab: 10mg/kg, iv,q3w Bevacizumab: 7.5mg/kg, iv, q3w HAIC: Oxaliplatin plus Fluorouracil/Leucovorin

SUMMARY:
To evaluate the efficacy and safety of HAIC combined with Cadonilimab and bevacizumab as first-line therapy in Unresectable hepatocellular carcinoma

DETAILED DESCRIPTION:
An open label, single-arm, single center, phase II study evaluating HAIC combined with cadonilimab and bevacizumab as first-line therapy in unresectable hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent signed prior to enrolment.
2. age 18-75 years, both sexes.
3. Histologically/cytologically confirmed HCC or cirrhosis meeting the clinical diagnostic criteria of HCC by American Association for the Study of Liver Diseases (AASLD).
4. ECOG PS of 0 or 1.
5. Absence of systemic anti-tumor treatment for HCC before the first dose.
6. Barcelona Clinic Liver Cancer (BCLC) stage of C. Stage B for those unsuitable for radical surgery and/or local treatment.
7. At least one measurable lesion according to RECIST V1.1, or measurable lesions showing definite progression following the local treatment based on RECIST V1.1.
8. Child-Pugh score of ≤ 7.
9. Sufficient organ and bone marrow functions, with the laboratory test values within 7 days before the enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other drugs via intravenous or subcutaneous administrations are allowed for correction treatment within the first 14 days after the laboratory test results are obtained). The specific information is as follows:

1) Routine blood test: absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 75 × 10^9/L; hemoglobin (HGB) ≥ 9.0 g/dL.

2) Hepatic function: total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN; serum albumin ≥ 28 g/L; alkaline phosphatase (ALP) ≤ 5 × ULN. 3) Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or clearance of creatinine (CCr) ≥ 50 mL/min (Cockcroft-Gault formula); urinalysis results showing urine protein <2+; patients whose baseline urinalysis results show urine protein ≥ 2+ should undergo 24-h urine collection and 24-h urine protein quantitation test result should be < 1 g.

4) Blood coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

10.Estimated survival ≥ 12 weeks. 11. Female patients of childbearing age or male patients with female sexual partners of childbearing age should take effective contraceptive measures throughout the treatment and 6 months after the last dose.

Exclusion Criteria:

1. Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma.
2. History of hepatic encephalopathy or liver transplantation.
3. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage.
4. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 104 copies/mL; hepatitis C virus (HCV) RNA > 103 copies/mL; hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive concurrently. Those who possess the indicators lower than the above criteria after nucleotide antiviral treatment can be enrolled.
5. Presence of metastasis to the central nervous system.
6. Presence of bleeding events from esophageal or gastric varices caused by portal hypertension within the past 6 months. Presence of known severe (G3) varicose vein in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator.
7. Presence of any life-threatening bleeding events within the past 3 months, including the need for transfusion, surgery or local treatment, and continuous medication therapy.
8. Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently. Presence of tumor thrombus of inferior vena cava.
9. A 10-day consecutive dosing of aspirin (> 325 mg/day) or other drugs, e.g., dipyridamole and clopidogrel, known to inhibit the platelet function within 2 weeks before the first dose.
10. History or current experience of pulmonary fibrosis and such lung diseases as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired lung function.
11. Uncontrolled/uncorrectable metabolic disorders, other non-malignant organ diseases, systemic diseases, or cancer-related secondary diseases with the potential to cause a relatively high medical risk and/or survival evaluation uncertainties unsuitable for subject enrollment as judged by the investigator; other circumstances unsuitable for subject enrollment as judged by the investigator.
12. Previous receipt of any antibody treatment involving anti-PD-1, anti-PD-L1/L2, or anti-CTLA4 or other immunotherapies. Previous receipt of anti-VEGF and/or VEGFR, RAF, MEK, PDGFR, and FGFR targeted therapy.
13. Pregnant or breastfeeding female patients.
14. lead to the following consequences: increased study participation or drug-related risks, or interference with interpreting trial results, and considered ineligible for participating in the trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) per RECIST 1.1 | Up to 1 year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Overall survival (OS) | Up to two years
  Defined as the time from enrollment to death from any cause
Progress Free Survival (PFS) | Up to two years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Adverse Events (AEs) | Up to two years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Disease Control Rate (DCR) per RECIST 1.1 | Up to 1 year
  Defined as proportion of patients who have CR or PR or SD

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No